CLINICAL TRIAL: NCT03135626
Title: Comparison of The Success Rates of Four Different Pulpotomy Techniques
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yeliz Guven, Dr, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/1728-1288
Record Dates: First submitted 2017-04-26; First posted 2017-05-01 (Actual); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Extensive Decay in Primary Molars
Keywords: Pulpotomy; Primary molars
MeSH Terms: interventions — tricalcium silicate; TheraCal; Pemetrexed; ferric sulfate

STUDY DESIGN:
Intervention Model Description: Split-mouth study design was used
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Biodentine (Experimental): Biodentine pulpotomy agent
  Interventions: Drug: Biodentine
- ProRoot MTA (Experimental): ProRoot MTA pulpotomy agent
  Interventions: Drug: ProRoot (Aggregate)
- MTA Plus (Experimental): MTA Plus pulpotomy agent
  Interventions: Drug: MTA Plus
- Ferric Sulfate 20% Dental Gel (Active Comparator): Ferric Sulfate %20 Dental Gel pulpotomy agent
  Interventions: Drug: Ferric Sulfate 20 % Dental Gel

INTERVENTIONS:
Drug: Biodentine
  Other Names: 77509635
  Arms: Biodentine
Drug: ProRoot (Aggregate)
  Other Names: 75896452
  Arms: ProRoot MTA
Drug: MTA Plus
  Other Names: 85303191
  Arms: MTA Plus
Drug: Ferric Sulfate 20 % Dental Gel
  Other Names: Viscostat
  Arms: Ferric Sulfate 20% Dental Gel

SUMMARY:
This randomized clinical trial was conducted to examine and compare the effectiveness of pulpotomy in primary molars treated with calcium silicate based materials including Biodentine and two different mineral trioxide aggregate (MTA) products (white ProRoot® MTA and MTA Plus®). Ferric sulfate pulpotomy was selected to represent the control group. 116 primary molars in 29 children were treated by pulpotomy and followed for a period of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients were eligible if they were 5 to 7 years old, healthy and cooperative, and had at least four carious primary molars, each of which was in a different quadrant and required a pulpotomy. The criteria for the selection of the teeth to be included in the study were presence of deep caries, presence of at least two-thirds of the root length radiographically and being restorable.

Exclusion Criteria:

* The exclusion criteria were the presence of any clinical or radiographic evidence of pulp degeneration (spontaneous or nocturnal tooth pain, tenderness to percussion, pathological mobility, internal or external root resorption, swelling or fistula, widened periodontal ligament (PDL) space, furcal or periapical radiolucency and teeth requiring more than 5 minutes to achieve hemostasis during clinical procedure. Teeth without permanent successor were not also included in the study.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2014-01-15 (Actual); Study Completion 2016-02-15 (Actual)

PRIMARY OUTCOMES:
Total success rate | 6 months after pulpotomy treatment
  Number of molars with both clinically and radiographically successful
Total success rate | 12 months after pulpotomy treatment
  Number of molars with both clinically and radiographically successful
Total success rate | 24 months after pulpotomy treatment
  Number of molars with both clinically and radiographically successful

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Guven, Dr., Principal Investigator — Istanbul University

IPD SHARING:
Plan to Share IPD: Undecided